CLINICAL TRIAL: NCT00501033
Title: A Prospective Comparative Study of Induction of Labor With a Cervical Ripening Double Balloon vs Foley Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Professor Jacob Bornstein, Western Galilee Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Induction of Labor; Cesarean; Endometritis
Keywords: Induction of labor; Cesarean; Endometritis; Foley; Infections
MeSH Terms: conditions — Endometritis; Infections | interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Mechanical induction of labor
Device: Double Balloon
Device: Foley Catheter

SUMMARY:
Hypothesis: The induction of labor in patients with unfavorable Bishop score is a challenging obstetrical process, and may be influenced or complicated by the cervical ripening method used. We will conduct a comparative study of the foley catheter vs the cervical ripening double balloon (Cook medical, GPN: G48149). We will compare the failure rates, cesarean section rate, infections and postpartum complications, especially endometritis.

DETAILED DESCRIPTION:
We will conduct a comparative study of the foley catheter vs the cervical ripening double balloon (Cook medical, GPN: G48149). We will compare the failure rates, cesarean section rate, infections and postpartum complications, especially endometritis. The study will include 200 parturients, 100 primiparous and 100 multiparous women. We will randomize each group to induction with the foley catheter or the cervical ripening double balloon. We will compare the failure rates, cesarean section rate, infectious and other postpartum complications, especially endometritis.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Parturients candidates for mechanical induction of labor

Exclusion Criteria:

* Suspected amnionitis
* Vaginal discharge
* Pre induction pyrexia
* Immunocompromised parturients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Success of labor induction | Postpartum period

SECONDARY OUTCOMES:
Postpartum endometritis rate | The postpartum period
Cesarean section rate | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ido Solt, MD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

REFERENCES:
- [Derived] Solt I, Frank Wolf M, Ben-Haroush S, Kaminskyi S, Ophir E, Bornstein J. Foley catheter versus cervical double balloon for labor induction: a prospective randomized study. J Matern Fetal Neonatal Med. 2021 Apr;34(7):1034-1041. doi: 10.1080/14767058.2019.1623776. Epub 2019 Jun 11. PMID 31185762